CLINICAL TRIAL: NCT02770456
Title: Fish Oil Supplementation to Prevent Preterm Delivery in China: A Randomized Controlled Trial
Brief Title: Fish Oil Supplementation to Pregnant Women in China
Acronym: FOPCHIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Fetal Programming, Denmark (Other)
Collaborators: Shanghai Institute of Planned Parenthood Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #6-FY01-317
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Premature Birth
Keywords: fish oil, preterm birth, pregnancy, China, prevention
MeSH Terms: conditions — Premature Birth | interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose fish oil (Experimental): Women will be offered 4 capsules per day containing fish oil
  Interventions: Dietary Supplement: High dose fish oil
- Low dose fish oil (Experimental): Women will be offered 4 capsules per day containing mixed fish oil and olive oil
  Interventions: Dietary Supplement: Low dose fish oil
- Control (Placebo Comparator): Women will be offered 4 capsules per day containing olive oil
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: High dose fish oil — Four 0.72-gram gelatine capsules per day with fish oil providing 2.0 g/d lc-n3FA
  Arms: High dose fish oil
Dietary Supplement: Low dose fish oil — Four 0.72-gram gelatine capsules per day with a mixture of fish oil and olive oil providing 0.5 g/d lc-n3FA
  Arms: Low dose fish oil
Dietary Supplement: Olive oil — Four 0.72-gram gelatine capsules per day with olive oil providing 0 g/d lc-n3FA
  Arms: Control

SUMMARY:
This randomized controlled trial with fish oil supplementation to pregnant women conducted in areas of China, which are generally low in fish intake and low income, aims at answering the following primary questions:

* Is a dose of 2.0 g/d long chain n-3 fatty acids efficient in preventing preterm birth
* Is a dose of 0.5 g/d long chain n-3 fatty acids efficient in preventing preterm birth
* Is a dose of 0.5 g/d as efficient as a dose of 2.0 g/d in affecting timing of spontaneous delivery in the preterm period

DETAILED DESCRIPTION:
The basic design is that of a randomized controlled trial with three groups randomized in ratios of 1:1:1. Two different doses of long chain n-3 fatty acids are tested against zero grams long chain n-3 fatty acids (lc-n3FA). These are provided in similarly looking gelatine capsules with either fish oil, a mixture (1:3) of fish oil and olive oil, or olive oil. Eligible women are randomized at around gestation weeks 16-24 and are asked to take the capsules until they have completed the preterm period (i.e. at 37 full gestation weeks) or until they deliver. Women are asked to complete questionnaires at randomization about diet and other baseline information, and again in gestation week 30 and after delivery. The trial is undertaken at hospitals in the two provinces of Gan-Su and Shaanxi. The three randomization groups will be compared with respect to proportions of preterm delivery. Cox regression will be used to compare the groups with respect to rates of spontaneous deliveries while accounting for elective delivery by regarding these as censoring events.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy without known complications

Exclusion Criteria:

* Regular user of fish oil
* Regular user of NSAIDs
* Known twin pregnancy

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5531 (Actual)
Dates: Start 2008-03; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Premature birth | 20 weeks on average, from randomization at gestation weeks 16-24 until on average gestation week 40
  Delivery occurring earlier than 259 gestation days

CONTACTS AND LOCATIONS:
Overall Officials: Sjurdur F Olsen, Ph.D., Study Director — Statens Serum Institut; Weijin Zhou, Ph.D., Principal Investigator — Shanghai Institute of Planned Parenthood Research

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Olsen SF, Halldorsson TI, Li M, Strom M, Mao Y, Che Y, Wang Y, Duan F, Olsen J, Zhou W. Examining the Effect of Fish Oil Supplementation in Chinese Pregnant Women on Gestation Duration and Risk of Preterm Delivery. J Nutr. 2019 Nov 1;149(11):1942-1951. doi: 10.1093/jn/nxz153. PMID 31387119